CLINICAL TRIAL: NCT05857514
Title: A Prospective, Open Label Randomized Controlled Trial of Prophylactic Rectal Indomethacin Versus Combined Pancreatic Duct Stent Placement and Rectal Indomethacin for Prevention of Post-ERCP Pancreatitis
Brief Title: Randomized Controlled Trial of Rectal Indomethacin Versus Combined Pancreatic Stent Placement and Rectal Indomethacin for Preventing Post-ERCP Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moti Lal Nehru Medical College (Other Government)
Responsible Party: Principal Investigator, Mukti Prakash Meher, Principal investigator, Moti Lal Nehru Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ECR/922/inst/UP/RR-2
Record Dates: First submitted 2023-04-09; First posted 2023-05-12 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Post-ERCP Acute Pancreatitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectal indomethacin (Active Comparator)
  Interventions: Drug: Rectal Indomethacin
- Pancreatic duct stent and rectal indomethacin (Active Comparator)
  Interventions: Procedure: Prophylactic Pancreatic duct stenting

INTERVENTIONS:
Drug: Rectal Indomethacin — Prophylactic Rectal indomethacin 100mg for prevention of post ERCP pancreatitis
  Arms: Rectal indomethacin
Procedure: Prophylactic Pancreatic duct stenting — Prophylactic pancreatic duct stenting with rectal indomethacin 100 mg for prevention of post-ERCP pancreatitis
  Other Names: Rectal indomethacin 100 mg
  Arms: Pancreatic duct stent and rectal indomethacin

SUMMARY:
The goal of this clinical trial is to compare rectal indomethacin alone versus combined pancreatic duct stenting and rectal indomethacin in prevention of post ERCP pancreatitis. The main question it aims to answer is: whether rectal indomethacin alone is superior to combination of pancreatic duct stenting and rectal indomethacin in prevention of post ERCP pancreatitis Participants will be patients who give consent to the study and who are required to undergo ERCP as part of their standard care.

If there is a comparison group: Researchers will compare [rectal indomethacin alone versus combined pancreatic duct stenting and rectal indomethacin in prevention of post ERCP pancreatitis.] to see if [whether rectal indomethacin alone is superior to combination of pancreatic duct stenting and rectal indomethacin in prevention of post ERCP pancreatitis].

ELIGIBILITY:
Inclusion Criteria:

1. Suspected sphincter of Oddi dysfunction
2. History of post ERCP Pancreatitis
3. Pancreatic instrumentation or sphincterotomy.
4. Precut sphincteroyomy
5. Difficult cannulation defined by more than 5 cannulation attempts
6. The use of double wire technique in bile duct access
7. At least 2 of the followings including

   1. Female age < 50 year
   2. 3 pancreatogram
   3. Acinarization (Contrast injection to tail of pancreas
   4. Normal serum bilirubin
   5. Guidewire to the tail of pancreas or secondary branches

Exclusion Criteria:

1. Patient planned for pancreatic stenting
2. Without informed consent
3. Age < 18 years
4. Pregnant women
5. Lactating women
6. Patient with altered anatomy
7. Contraindications to the use of NSAIDS
8. Renal failure
9. Ongoing or recent hospitalisation for acute pancreatitis
10. Allergy to aspirin or NSAIDs
11. known chronic calcific pancreatitis -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
To compare rectal indomethacin alone versus combined pancreatic duct stent and rectal indomethacin in prevention of post ERCP pancreatitis | 24 hour
  For comparison between these two arms the investigators will measure serum amylase in U/L value after 6 hour and 24 hour of the ERCP procedure. The investigators will also assess for pain abdomen and vomiting suggestive of acute pancreatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Mukti Pr Meher, MBBS, MD, Principal Investigator — Investigator
Locations (2):
- India (2):
  - Department of Gastroenterology and Hepatology, MLN Medical college and SRN Hospital, Allahābād, Uttar Pradesh
  - Department of Gastroenterology and Hepatology, Allahābād, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No